CLINICAL TRIAL: NCT05958329
Title: Remote Short Sessions of Heart Rate Variability Biofeedback
Brief Title: Short Sessions of HRV Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robert Hirten, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-00596
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Resilience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRV Biofeedback (Experimental): 5 minute daily sessions of HRV biofeedback
  Interventions: Behavioral: HRV Biofeedback

INTERVENTIONS:
Behavioral: HRV Biofeedback — 5 minute daily sessions of HRV biofeedback

SUMMARY:
Remote 5 minute sessions of heart rate variability (HRV) biofeedback will be employed by participants for 5 weeks. Subjects will be followed for a total of 17 weeks. Surveys assessing psychological well being will be completed during the study period. Wearable devices will be worn to monitor HRV response during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Participants were recruited from The Mount Sinai Hospital, Morningside Hospital, Mount Sinai West, Mount Sinai Beth Israel, Mount Sinai Queens, New York Eye and Ear Infirmary, and Mount Sinai Brooklyn.
* Eligible participants were 18 years of age or greater.
* Had an iPhone series 5 or greater.
* Had or were willing to wear an Apple Watch 4 or greater.
* Potential participants were excluded if they had an underlying chronic disease or used a medication that is known to impact autonomic nervous system function.

Exclusion Criteria:

* Underlying chronic diseases including but not limited to:

  * rheumatoid arthritis
  * systemic lupus erythematosus
  * inflammatory bowel disease
* Use of medications that impact heart rate variability including but not limited to:

  * beta-blockers (ie. atenolol, carvedilol, metoprolol, Coreg, Tenormin, Normodyne, Trandate)
  * digoxin
  * calcium channel blockers (ie. Norvasc, amlodipine, Cardene, nicardipine, Procardia, nifedipine, Cardizem, diltiazem)
  * regularly used benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Up to Week 7
  Heart rate variability measured in milliseconds (ms) at 7 weeks compared to baseline. Higher rates indicate increased parasympathetic nervous system activity.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC | Up to Week 17
  Resilience: the Connor-Davidson Resilience scale (CD-RISC) quantifies stress coping ability. The CD-RISC is a 25-item self-administered scale. Scoring of the full 25 item scale is based on summing the total of each item, which is scored from 0-4. The full range is therefore from 0 to 100, with higher scores reflecting greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hirten, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Health care worker data is included in the dataset.